CLINICAL TRIAL: NCT01780948
Title: Drug Interaction and Pharmacokinetic Assessment of Everolimus When Coadministered With Atorvastatin in Renal Transplantation Recipient
Brief Title: Pharmacokinetic of Everolimus and Atorvastatin Co-administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Ratchadapiseksompotch Research Fund (Unknown)
Responsible Party: Principal Investigator, ANOCHA WANITCHANONT, Department of Medicine, Faculty of Medicine, Chulalongkorn University, Chulalongkorn University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A7478
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Difference of 12-hour AUC
Keywords: Drug Interaction; Pharmacokinetics; Everolimus; Atorvastatin
MeSH Terms: interventions — Atorvastatin; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- everolimus (Placebo Comparator): Everolimus administration with adjusted dose to target C trough (C0) level between 3-12 ng/mL
  Interventions: Drug: Atorvastatin 20 mg
- everolimus with atorvastatin 20 mg (Experimental): Co-administration of everolimus and atorvastatin. Everolimus administration with adjusted dose to target C trough (C0)level between 3-12 ng/mL.
  Atorvastatin 20 mg/day (fixed dose)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Atorvastatin 20 mg — Add atorvastatin 20 mg and compare 12-hour AUC of everolimus between Arm everolimus and everolimus with atorvastatin 20 mg
  Other Names: Lipitor 20 mg
  Arms: everolimus
Drug: Everolimus — Administration only everolimus, no atorvastatin. Everolimus administration with adjusted dose to target C trough (C0)level between 3-12 ng/mL.
  Other Names: Everolimus alone
  Arms: everolimus with atorvastatin 20 mg

SUMMARY:
Hypothesis : In renal transplantation recipient who received immunosuppressive drug "certican" and have hypercholesterolemia will get lipid lower drug-HMG Co-A reductase inhibitors. Because atorvastatin and everolimus have metabolism via Cytochrome P450 subfamily 3A4 both, so investigator made the hypothesis that when patients received everolimus with atorvastatin will change area under the time concentration curve of everolimus.

DETAILED DESCRIPTION:
Population : Thai postrenal transplantation recipient who received everolimus and have hypercholesterolemia in posttransplantation clinic at Faculty of Medicine, Chulalongkorn University.

Study Design : Experimental study, Two-sample crossover study Sample size calculation :N = 18 Primary outcome : 12-hour area under the time concentration curve of everolimus Secondary outcome : renal function (serum creatinine, creatinine clearance)

Method :

1. Patients will random to everolimus or everolimus with atorvastatin 20 mg arm for 1 month.
2. Take blood sample for everolimus concentration at time 0,0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 hour
3. After first blood sample, patients will received everolimus only for 1 month (wash out period)
4. Patients will switch to another arm eg.patient who had received everolimus will switch to everolimus with atorvastatin 20 mg for 1 month
5. Take blood sample for everolimus concentration at time 0,0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 hour
6. Everolimus level will analyse for 12-hour AUC of everolimus.

ELIGIBILITY:
Inclusion Criteria:

* Post renal transplantation recipient who received immunosuppressive drug Everolimus and has hypercholesterolemia
* Co everolimus level within 3-12 ng/mL
* Informed consent
* Patient can follow research methodology

Exclusion Criteria:

* Patient don't want to participate in the study
* Post renal transplantation recipient who have normal lipid profile

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
12-hour area under the time concentration curve of everolimus | 3 months
  compare when taking only everolimus to coadministered with atorvastatin

SECONDARY OUTCOMES:
Renal function | 3 months
  Renal function : serum creatinine, 24 hour creatinine clearance 24 hour urine protein, Urinalysis Sample take at month 0,1,2,3
Liver function test | 3 month
  Total protein, Albumin, total bilirubin, direct bilirubin, AST, ALT, Alkaline phosphatase at month 0,1,2,3
Lipid profile | 3 month
  Total cholesterol, Triglyceride, HDL, LDL at month 0,1,2,3
Rhabdomyolysis | 3 month
  Adverse drug reaction from atorvastatin by measured CPK at month 0,1,2,3

OTHER OUTCOMES:
Correlation of 12-hour AUC and point of everolimus level | 3 months
  To correlate between 12-hour AUC and point of everolimus level

CONTACTS AND LOCATIONS:
Overall Officials: Anocha Wanitchanont, MD., Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Kovarik JM, Hartmann S, Hubert M, Berthier S, Schneider W, Rosenkranz B, Rordorf C. Pharmacokinetic and pharmacodynamic assessments of HMG-CoA reductase inhibitors when coadministered with everolimus. J Clin Pharmacol. 2002 Feb;42(2):222-8. doi: 10.1177/00912700222011148. PMID 11831546